CLINICAL TRIAL: NCT05390008
Title: The Effects of Pelvic Floor Muscle Training and Modified Pilates Exercises in Elderly Women With Stress Urinary Incontinence
Brief Title: The Effects of PFMT and MPE in Elderly Women With SUI.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ebru Kaya Mutlu, PT, Assoc. Prof., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06/05/2022
Record Dates: First submitted 2022-05-18; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Stress Urinary Incontinence; Pelvic Floor Disorders; Aging
Keywords: aging; exercise; pelvic floor; urinary incontinence; women
MeSH Terms: conditions — Urinary Incontinence, Stress; Pelvic Floor Disorders; Motor Activity; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Pelvic Floor Muscle Training (Experimental): volunteer elderly women with SUI
  Interventions: Other: Pelvic Floor Muscle Training
- Group 2: Modified Pilates Exercises (Experimental): volunteer elderly women with SUI
  Interventions: Other: Modified Pilates Exercise

INTERVENTIONS:
Other: Pelvic Floor Muscle Training — In order to increase participants' PFM strength and endurance , PFMT was taught two days a week for 12 weeks. This training included two type of exercises that consisted of fast and slow PFM contractions.
  Fast Contractions: This exercise was done in sitting position, While participants' arms were on thighs with their feet resting on the floor and sitting unsupported on the back of their seat. They were taught how to quickly contract and relax their PFM.
  Slow Contractions: The practice position of this exercise was in sitting position as it happened in fast contraction. This training lasted for 12 weeks and it was divided into periods as 1-3 week, 4-6 week, 7-9 week, 10-12 week. In the forth coming weeks of this period, the number of exercise repetitions and the number of sets were increased.
  Arms: Group 1: Pelvic Floor Muscle Training
Other: Modified Pilates Exercise — Before starting the 12-week practice protocol, the concept of stabilization was explained to the participants. Participants were taught how to control the core region by using the stabilizer device and the basic principles of pilates. The exercise program was planned that would last 50 minutes. This program was carried out as three-stage and these stages were warm-up phase, main exercise program and cool down phase. The allocated times for the warm-up phase was 10 minutes. The allocated time for the main exercise program was 30 minutes and active resting was done by performing breathing exercises in the 15th minute of the main exercise program. The allocated time for the cool down phase was 10 minutes. Each exercise was done as 10 repetitions then the next exercise was started.
  The exercises of the second 6 weeks were performed by adding a red elastic exercise band at the beginner-intermediate level, which released 1.7 kg force with 100% stretching.
  Arms: Group 2: Modified Pilates Exercises

SUMMARY:
The aim of the study was to compare the effects of PFMT and MPE on SUI frequency and explosure from symptoms, PFM activation response and strength of lumbar stabilizing muscle in elderly women with SUI.

DETAILED DESCRIPTION:
Stress Urinary Incontinence (SUI) is associated with situations which bladder pressure exceeds the pressure at which the urethra has the capacity to remain closed, such as physical exertion, coughing, and sneezing. SUI is more predominant in women worldwide, with a prevalence ranging from 10% in young women to 45% in the elderly. Physiotherapy interventions in SUI include patient education including recommendations for bladder and/or bowel training, fluid management, and diet modification; modalities for decrease pain; pelvic floor muscle training (PFMT) with or without biofeedback and/or electrical stimulation to improve strength and coordination of the pelvic floor muscle (PFM) and stabilization exercises to improve strength of abdominal and/or lumbar stabilizer muscles.

PFMT includes repetitive contraction of the PFM, which increases perineal support and improves the muscle tone of the PFM. Modified pilates exercises (MPE) is a mind-body approach that includes slow, controlled movements that focus on posture and breathing.

The aim of the study was to compare the effects of PFMT and MPE on SUI frequency and explosure from symptoms, PFM activation response and strength of lumbar stabilizing muscle in elderly women with SUI. In this study, thirty-four elderly women who were diagnosed with SUI were randomized into Group 1: PFMT (n=17) or Group 2: MPE (n=17). Both groups performed their exercises twice a week for 12 weeks and accompanied by a physiotherapist. Incontinence Severity Index (ISI), Urogenital Distress Inventory-Short Form (UDI-6) and Incontinence Impact Questionnaire-Short Form (IIQ-7) were used to assess SUI frequency and explosure from symptoms, electromyography (EMG) device was used to assess PFM activation response and a stabilizer was used to assess strength of lumbar stabilizing muscle. The assessments were performed at baseline and after 12 week treatment. The effect size was calculated for the assessments used in the study.

ELIGIBILITY:
Inclusion Criteria:

1. being volunteer to participate in a study;
2. being a woman over the age of 65;
3. having the diagnosis of SUI;
4. participants who scored at least 24 on the Mini Mental State Exam (MMSE).

Exclusion Criteria:

1. having a neurological disease;
2. having PFM which cannot contract;
3. having a urinary tract infection;
4. having the stage two or higher pelvic organ prolapse; and
5. participants who received a SUI treatment in the recent year.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Elderly women
Enrollment: 30 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
SUI frequency change - Incontinence Severity Index (ISI) | SUI frequency was assessed by Incontinence Severity Index (ISI) at before and after 12 weeks of treatment
  Incontinence Severity Index (ISI) was used to determine the UI frequency of the participants. This test consisted of two questions, regarding frequency and amount of leakage. Incontinence severity was determined by multiplying assigned values of two questions' responses. By taking into account the results, urine leakage was identified according to the following scale; 1-2 as 'slight', 3-4 as 'moderate', 8-9 as 'severe', 12 as 'very severe'.
SUI frequency and explosure from symptoms change - Urogenital Distress Inventory-Short Form (UDI-6) | SUI frequency and explosure from symptoms was assessed by Urogenital Distress Inventory-Short Form (UDI-6) at before and after 12 weeks of treatment
  Urogenital Distress Inventory-Short Form (UDI-6) questionnaire was used to measure the participants' exposure to incontinence symptoms. In this form consisting of 6 questions, each question takes values in the range of 0-4. Then, the total value is converted to values ranging from 0-100. A score of 0 indicates that the patient is not bothered at all, while a score of 100 indicates that the patient is extremely disturbed by this symptom.
SUI frequency and explosure from symptoms change - Incontinence Impact Questionnaire-Short Form (IIQ-7) | SUI frequency and explosure from symptoms was assessed by Incontinence Impact Questionnaire-Short Form (IIQ-7) at before and after 12 weeks of treatment
  Incontinence Impact Questionnaire-Short Form (IIQ-7) was used to determine the extent to which urinary symptoms affect the participants' activities of daily living, social relationships and psychological states. This form included 7 questions and each question was assigned a value from 0 to 3. Then, the total value is converted to values ranging from 0-100. A score of 0 indicates that the patient is not bothered at all, while a score of 100 indicates that the patient is extremely disturbed by this symptom.
PFM activation change - MyoPlus4Puro-EMG device | PFM activation was assessed by MyoPlus4Puro-EMG device at before and after 12 weeks of treatment
  MyoPlus4Puro-EMG device was used to determined the participants' PFM activation. The measurement was performed while subjects' knees were positioned at 140° of flexion with soles in the bed and there was a 30 cm gap between the feet. Active electrodes were placed on the right and left side of the perineal body. Passive electrode was located in front of the femoral. The length of contraction lasted five seconds and resting lasted five seconds, too. Five repeated contractions with a five second pause between each contraction were performed in total and the measurement lasted 50 seconds. However, in order for the contraction to be only in the pelvic floor muscles, before the measurement, the subjects were told how to perform the correct pelvic floor contraction without contracting the abdominal, hip and thigh muscles and without holding the breath.
Strength of lumbar stabilizing muscle change - Stabilizer Pressure Biofeedback | Strength of lumbar stabilizing muscle was assessed by stabilizer at before and after 12 weeks of treatment
  Stabilizer Pressure Biofeedback device was used to determine the strength of lumbar stabilizing muscle. Subjects were asked to be in the face-down position and the pillow was located in the abdominal region. The bottom edge of the pillow was placed in paralel with crista iliaca. Meanwhile, subjects' knees were in flat position, arms were by their side and their head was in a relaxed position. After the manometric pressure was adjusted to 70 mmHg, participant was asked to slowly contract his/her transversus abdominis (TrA) muscle. That's why, subject was instructed by saying 'suck your belly in'. The decrease of pressure value increases in direct proportion to the to the magnitude of the stabilization force. Three tests were completed in total and the average value was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Kaya Mutlu, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Darulaceze Directorate of Istanbul, Istanbul, Kayisdagi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Falah-Hassani K, Reeves J, Shiri R, Hickling D, McLean L. The pathophysiology of stress urinary incontinence: a systematic review and meta-analysis. Int Urogynecol J. 2021 Mar;32(3):501-552. doi: 10.1007/s00192-020-04622-9. Epub 2021 Jan 8. PMID 33416968
- [Background] Oliveira M, Ferreira M, Azevedo MJ, Firmino-Machado J, Santos PC. Pelvic floor muscle training protocol for stress urinary incontinence in women: A systematic review. Rev Assoc Med Bras (1992). 2017 Jul;63(7):642-650. doi: 10.1590/1806-9282.63.07.642. PMID 28977091
- [Background] Celiker Tosun O, Kaya Mutlu E, Ergenoglu AM, Yeniel AO, Tosun G, Malkoc M, Askar N, Itil IM. Does pelvic floor muscle training abolish symptoms of urinary incontinence? A randomized controlled trial. Clin Rehabil. 2015 Jun;29(6):525-37. doi: 10.1177/0269215514546768. Epub 2014 Aug 20. PMID 25142280
- [Background] Lausen A, Marsland L, Head S, Jackson J, Lausen B. Modified Pilates as an adjunct to standard physiotherapy care for urinary incontinence: a mixed methods pilot for a randomised controlled trial. BMC Womens Health. 2018 Jan 12;18(1):16. doi: 10.1186/s12905-017-0503-y. PMID 29329567
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322